CLINICAL TRIAL: NCT03221673
Title: Relationship of Physical Activity and Diet With Socio-demographic, Environmental, and Metabolic Factors in Arkansas Public School Children
Brief Title: Arkansas Active Kids! -Objective 3
Acronym: AAK
Status: Completed | Type: Observational
Sponsor: Arkansas Children's Hospital Research Institute (Other)
Collaborators: USDA Beltsville Human Nutrition Research Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Elisabet Borsheim, Associate Professor, Arkansas Children's Hospital Research Institute
Other Study IDs: 3092-51000-056-04A
Record Dates: First submitted 2017-06-28; First posted 2017-07-18 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Physical Activity; Child
Keywords: Exercise; Children; Arkansas; Physical activity; Sedentary
MeSH Terms: conditions — Motor Activity; Sedentary Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Whole blood, serum, stool, saliva, urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a cross-sectional study aiming to identify how daily activities affect children's body fitness and general health. Also, the study will address how specific behaviors (such as diet and sleep) as well as neighborhood and home environment affect children's metabolic health and fitness level.

DETAILED DESCRIPTION:
The purpose of this study is to determine how daily activities, home, neighborhood and school environments affect Arkansas children's health. Children from Central Arkansas ages 7-10 years will be recruited to participate in a variety of physical activity tests including strength, flexibility, balance and endurance. During these tests, participants will perform tasks such as cycling on a stationary bike and extending and flexing their knees on a special type of chair. Body composition will be measured and blood, saliva, urine and stool samples collected. Participants and parents will be asked to complete questionnaires on physical activity, home and neighborhood environment as well as sleeping habits. Finally, participants will wear an accelerometer based monitor that will track their physical activity and sleeping patterns. One in person visit will take place at Arkansas Children's Nutrition Center (Little Rock, AR) and will last up to 8 hours. Reimbursement will be provided.

ELIGIBILITY:
Inclusion Criteria:

* Ages 7 to 10 years
* Boys or girls
* All ethnicities
* All BMIs (all body types)

Exclusion Criteria:

* Severe persistent asthma (determined by daily use of oral/inhaled corticosteroid to keep asthma symptoms under control and/or frequent use of rescue inhaler)
* Type 2 diabetes mellitus
* Other pre-existing medical conditions or medications as determined by the investigators to affect the outcomes of interest

Ages: 7 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Up to 300 pre-pubertal children ages 7 to 10 years old, both boys and girls, will be recruited from Central Arkansas.
Sampling Method: Non-Probability Sample
Enrollment: 230 (Actual)
Dates: Start 2017-05-18 (Actual); Primary Completion 2018-09-25 (Actual); Study Completion 2018-09-25 (Actual)

PRIMARY OUTCOMES:
Correlation between fitness level and metabolic health | June 2016-August 2018
  A fitness test will be performed to determine peak oxygen uptake (VO2 peak, ml/kg per min). Correlations between peak VO2 and different markers of cardiometabolic health (IL-6, triglycerides, non-esterified fatty acids, glucose, insulin concentrations, etc.) will be determined. Other indicators of fitness level such as strength, flexibility and balance will be measured and correlations assessed.

SECONDARY OUTCOMES:
Correlation between home and neighborhood environments and fitness level | June 2016-August 2018
  Home and neighborhood environments will be assessed via interviewer administered questionnaires. Scores obtained from these questionnaires will be correlated with peak oxygen consumption, strength, flexibility and balance scores.

CONTACTS AND LOCATIONS:
Overall Officials: Elisabet Borsheim, Ph.D., Principal Investigator — Arkansas Children's Nutrition Center and Arkansas Children's Research Institute
Locations (1):
- Arkansas Children's Nutrition Center, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared with researchers outside the study.

REFERENCES:
- See also: Arkansas Children's Nutrition Center webpage — https://medicine.uams.edu/pediatrics/research/acnc/